CLINICAL TRIAL: NCT04156217
Title: A Pilot Study of EBV-TCR-T Cells in EB Virus Infection Diseases After HSCT
Brief Title: EBV-TCR-T Cells for EB Virus Infection After HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-004
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-08

CONDITIONS: EBV Emia and EBV Positive PTLD After Allogenic HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-TCR-T cells (Experimental): Patients with EBV emias or EBV positive PTLD will be enrolled, and donor derived EBV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.1-1×106 EBV-TCR-T cells. The EBV DNA copies and EBV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28).
  Interventions: Biological: EBV-TCR-T cells

INTERVENTIONS:
Biological: EBV-TCR-T cells — EBV-TCR-T cells are prepared via lentiviral infection. patients with EBV emias or EBV positive PTLD will be enrolled, and donor derived EBV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.1-1×106 EBV-TCR-T cells. The EBV DNA copies and EBV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28).

SUMMARY:
This is a single center, single arm, open-label, phase I study to evaluate the safety and efficacy of EBV-TCR-T cells in patients with EB virus infection after HSCT.

DETAILED DESCRIPTION:
EBV infection is a common virus infection of HSCT, and which is highly related with the failure of transplantation and survival time of transplant patients. To evaluate the safety and efficacy of allogenic EBV-TCR-T cell therapy in subjects with EBV infection, patients with EBV emias or EBV positive PTLD will be enrolled, and donor derived EBV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.1-1×106 EBV-TCR-T cells. The EBV DNA copies and EBV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28).

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-70 years, including boundary values, gender unlimited;
2. The EBV DNA copies number of allogenic HSCT patients with EBV infection (EBV emia and EBV positive PTLD) still did not decrease，after treated with lower dosage of Immunosuppressants，or antiviral therapy or Rituximab（Rituxan）；
3. Allogenic HSCT patients could not tolerate the antiviral therapy and / or Rituximab（Rituxan）；
4. The EBV-positive diagnosis criteria: EBV DNA copy number>1000 copies/ ml, or the tissue EBV-EBER pathological result is positive, the diagnosis of PTLD was based on the diagnostic criteria of WHO 2016；
5. Estimated life expectancy ≥ 3 months；
6. ECOG 3 ；
7. Patients who voluntarily sign informed consent and are willing to comply with treatment plans, visit arrangements, laboratory tests and other research procedures.

Exclusion Criteria:

1. Patients with active aGVHD III-IV and / or mild and severe cGVHD;
2. Received cell therapy such as DLI,CTL,CAR-T or participated in any other clinical study of drugs and medical devices before 30 days of enrollment；
3. Pregnant or lactating women;
4. Intracranial hypertension or confusion; respiratory failure; disseminated intravascular coagulation;
5. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability;
6. The researchers found that it was unsuitable for the recipients to be enrolled.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of adverse events | 3months
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Proliferation ratio of TCR-T cells | 3months
changes of EBV-DNA copies | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China